CLINICAL TRIAL: NCT07178132
Title: Comparative Effects of Tissue Flossing and Proprioceptive Neuromuscular Facilitation on Hamstring Flexibility and Knee Range of Motion in Young Female Students
Brief Title: Use of PNF and Tissue Flossing to Treat Hamstring Tightness in Young Female Students
Acronym: Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakshi Negi (Other)
Collaborators: Guru Nanak Dev University (Other)
Responsible Party: Sponsor-Investigator, Sakshi Negi, Principal Investigator, Guru Nanak Dev University
Organization: Guru Nanak Dev University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2250/HG
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hamstring Tightness; Muscle Tightness
Keywords: tightness; tissue flossing; proprioceptive neuromuscular facilitation; Hamstring tightness; flexibility
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue Flossing Arm (Experimental): Application of tissue floss band to hamstring muscle at moderate tension for 2 minutes, followed by flexibility testing via AKET (Active Knee Extension Test), PKET (Passive Knee Extension Test), SLR (Straight Leg Raise), and Sit-and-Reach.
  Interventions: Other: tissue floss band
- PNF Hold-Relax Arm (Active Comparator): Standard PNF hold-relax stretching technique of hamstring, followed by flexibility testing via AKET (Active Knee Extension Test), PKET (Passive Knee Extension Test), SLR (Straight Leg Raise), and Sit-and-Reach.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: tissue floss band — Floss band is wrapped in thigh from distal to proximal for 2 minutes. during this period patient is asked to actively perform movement for 2 minute, after that the band is removed and repeated once more. Immediately followed by flexibility measurements
  Other Names: Floss band
  Arms: Tissue Flossing Arm
Other: Proprioceptive Neuromuscular Facilitation — Proprioceptive Neuromuscular Facilitation (PNF) Stretching using the hold-relax method: participants perform an isometric contraction of the hamstring at the end of its stretch range , followed by relaxation and passive stretch, then flexibility assessed similarly
  Arms: PNF Hold-Relax Arm

SUMMARY:
The goal of this clinical trial is to learn tissue flossing and proprioceptive neuromuscular facilitation effect in treating hamstring muscle tightness.

The main questions it aims to answer are:

1. which technique is more useful in giving instant relaxation of hamstring muscle
2. can these technique increase muscle flexibility and knee motion

Researchers will compare Tissue flossing to a PNF (Proprioceptive neuromuscular facilitation) to see which on is more effective.

Participant will:

1. be provided one technique either tissue flossing or PNF in first day
2. physiotherapist will immediately measure the the change in flexibility or knee motion

2. another technique will be applied after 1 week 3. again change in flexibility and knee motion will be recorded

ELIGIBILITY:
Inclusion Criteria:

* Female subjects were included in the study
* Subjects with hamstring muscle tightness were included
* Subjects between the age group of 18-25 years were included

Exclusion Criteria:

* Male subjects
* Subject who didn't fulfill the age criteria
* Subject with hamstring tear or other knee ligament injury
* Any history of lower limb surgery dating back a year
* Subjects with Lower back pain or any neurological compromise in the lower limb
* Any acute injury like a sprain, strain, and open wound
* Subjects who had latex allergies
* Subjects with venous thrombotic disease, heart disease, respiratory illness, and dermatitis, in their lower legs were excluded

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants were eligible for inclusion in this study. The study focused on young women because sex-related differences in hamstring flexibility, joint range of motion, and neuromuscular properties have been reported in the literature. Restricting the sample to female students provided a more homogeneous group and reduced variability related to gender differences, thereby enhancing internal validity
Enrollment: 60 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Active Knee Extension Test | From enrollment to the end of treatment at 1 week
  With the participant supine and the hip flexed to 90°, the participant actively extends the knee. A goniometer was used to records the knee extension angle. Three trials are performed and the mean is used for analysis.
Passive Knee Extension Test | From enrollment to the end of treatment at 1 week
  With the participant supine and the hip flexed to 90°, the examiner passively extends the knee until the first onset of resistance. A goniometer is used to records the knee extension angle. Three trials are performed and the mean is used.
Straight Leg Raise | From enrollment to the end of treatment at 1 week
  With the participant supine, the examiner passively raises the extended leg until resistance . A goniometer at the hip measures maximum hip flexion angle (degrees). Three trials are performed and the mean is used.
Sit-and-Reach Test | From enrollment to the end of treatment at 1 week
  The participant sits with legs extended and reaches forward along a standard sit-and-reach box . After a warm-up, three trials are performed and the mean score (cm) is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet Kaur, MPT, Study Director — Guru Nanak Dev University
Locations (1):
- Guru Nanak Dev University, Amritsar, Punjab, India

IPD SHARING:
Plan to Share IPD: No
I did not include individual participant data in ClinicalTrials.gov to protect participant privacy and confidentiality.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT07178132/Prot_SAP_000.pdf